CLINICAL TRIAL: NCT04500639
Title: Do Common Medications Alter the Course of COVID-19?
Brief Title: Over-the-counter Medications & COVID-19
Acronym: OTC℞&COVID19
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100243
Record Dates: First submitted 2020-08-04; First posted 2020-08-05 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2 Infection; Covid19
Keywords: Ibuprofen; Over-the-counter medications
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ibuprofen is one of several common medications implicated in coronavirus disease 2019 (COVID-19) severity. On March 11, the Lancet Respiratory Medicine published a letter stating ibuprofen can increase angiotensin-converting enzyme 2 (ACE2) expression. On March 14, the French Minister of Health tweeted that ibuprofen should be avoided because it will aggravate COVID-19. This concern was echoed by scientists and senior doctors in the British Medical Journal news on March 17. In response, the World Health Organization (WHO) issued a recommendation on March 18 to avoid ibuprofen in people with symptoms of COVID-19. However, the WHO reversed this recommendation the next day because of insufficient evidence. Health Canada issued a safety alert on March 20 stating there was no evidence that ibuprofen worsens COVID-19 symptoms. There is some evidence suggesting NSAID use (primarily ibuprofen) can increase severity of community acquired bacterial pneumonia in hospitalized children and adults. However, we do not know if ibuprofen use alters the course of COVID-19.

Ibuprofen is an effective analgesic and antipyretic medication. People often use over-the-counter cough and cold products containing ibuprofen to manage symptoms of a respiratory tract infection before they seek medical attention. Therefore, exposure to ibuprofen is highly probable in people with COVID-19 symptoms. Patients, clinicians, and policy makers need to know if ibuprofen is safe to use in management of COVID-19 symptoms.

This case-control study will explore the association between common medications and COVID-19 severity in a cohort of people tested for SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the province of Alberta tested for COVID-19 since March 1, 2020

Exclusion Criteria:

* Individuals who are currently hospitalized, who died, or who do not have contact information in the COVID-19 test record

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Albertans seeking testing for COVID-19 are eligible for inclusion in the study. Invitation letters will be sent to all individuals with positive test results and a random sample of individuals with negative test results.
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Ibuprofen exposure for symptom management | Prior to COVID-19 testing
  Ibuprofen use will be determined from responses to a survey question asking what over-the-counter medications were used to help manage symptoms before testing for COVID-19. Response options include all brand name analgesic and cough and cold products available in Canada, as well as options to list generic brand products containing ibuprofen or acetaminophen.
  If a participant indicates they used both acetaminophen and ibuprofen to manage symptoms, an additional question will ask for the sequence that these analgesics were started. Responses to this question will help us determine if ibuprofen was added for better symptom relief, presumably because symptoms were severe.

SECONDARY OUTCOMES:
Exposure to other drugs implicated in COVID-19 severity | Prior to COVID-19 testing
  Exposure to angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs), mineralocorticoid receptor antagonists (MRAs), and pioglitazone will be identified using additional questions in the survey and verified with prescription drug records in the administrative health databases.

CONTACTS AND LOCATIONS:
Overall Officials: Scot Simpson, PharmD, MSc, Principal Investigator — Faculty of Pharmacy and Pharmaceutical Sciences, University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
A data management plan will be posted on https://portagenetwork.ca/ when it is available.